CLINICAL TRIAL: NCT02492347
Title: Is Antenatal Exposure to Selective Serotonin Reuptake Inhibitors (SSRIs) Associated With Prolongation of the QT Interval in Term Neonates (Greater Than 37 Complete Weeks Gestation)?
Brief Title: Effect of Antenatal SSRI Exposure on the QT Interval of Neonates
Acronym: SSRIs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southampton (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 8442
Record Dates: First submitted 2015-06-17; First posted 2015-07-08 (Estimated); Last update posted 2017-11-06 (Actual); Status verified 2017-11

CONDITIONS: Qt Interval, Variation in; Adverse Effect of Selective Serotonin Reuptake Inhibitors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Neonates exposed to AN SSRI use (Active Comparator): A group of newborn babies who have been exposed to SSRIs in pregnancy will receive an Electrocardiogram at 48-72 hours of age.
  Interventions: Procedure: Electrocardiogram
- Neonates not exposed to AN SSRI use (Other): A group of newborn babies, who require treatment with intravenous antibiotics for at least 36 hours, having been identified as being at risk of having an infection within 12 hours of being born. They are subsequently confirmed as clinically well and will receive an Electrocardiogram at 48-72 hours of age.
  Interventions: Procedure: Electrocardiogram

INTERVENTIONS:
Procedure: Electrocardiogram — The ECG is a non-invasive screening tool. It will be performed when the neonate is settled and comfortable. The electrodes used are made with soft jelly adhesive which is stored at room temperature. The procedure will be conducted in a timely manner, taking no longer than 15 minutes. The electrodes are easily removed, and the neonate redressed.

SUMMARY:
Selective Serotonin Reuptake Inhibitors (SSRIs) are a group of antidepressants that suppress the re-absorption of a chemical called Serotonin in the brain, and improve mood. SSRI use in the treatment of mental health problems has increased greatly since their introduction in the 1980's. When given in pregnancy they cause less fetal effects than other antidepressants. However they are still known to cause premature birth, heart defects and withdrawal symptoms in the baby. Withdrawal symptoms can occur in up to 30% of exposed babies, where as heart defects have been found to increase by 2-3 times against the normal rate of 1%. There is very limited information available, but it is also thought it may cause lengthening of a certain portion of the heart beat, the QT interval, which has been shown to lead to sudden death in adults. The QT interval will be looked at in this study, comparing babies exposed to SSRIs in pregnancy with unexposed babies.

The study will be based in the United Kingdom (UK), at the Maternity Unit of a District General Hospital, and will be carried out over 12-18 months.

A group of babies whose mothers took SSRIs whilst pregnant will have an Electrocardiogram (ECG) done when they are 2-3 days old. These will be compared with babies whose mothers did not, but whose babies were still in hospital because they were at risk of having an infection, but were found to be healthy.

The study hopes to see whether there is a link between SSRI use in pregnancy and lengthening of the QT interval and if so, extra surveillance may be considered for this group of babies.

DETAILED DESCRIPTION:
The study will be carried out at the maternity unit of the local district general hospital. It is normal practice for women who have taken SSRIs in pregnancy to deliver at the local district general hospital, rather than at home or in the community, due to the possible problems with their babies.

Currently it is standard practice for a plan of care for after the baby is born (an ALERT) to be generated whilst the woman is pregnant. The ALERT form is developed by specialist nurses, Advanced Neonatal Nurse Practitioners (ANNPs) and Doctors specialising in newborn babies. The ALERT form details the recommended place of birth; length of expected hospital stay; known side effects of SSRIs; the monitoring that is done after birth and why; and whether breastfeeding is advised. This is returned to community midwifery staff to discuss with the woman ahead of delivery. When the woman who has taken SSRIs in her pregnancy comes to the maternity unit to deliver the ALERT form is activated. After birth she will be assessed by maternity staff and ANNPs to see if her baby is suitable for the study, and if so, she will be given an information leaflet and invitation letter when her baby is 12 hours old by these staff.

The other group of mothers that will be asked for the participation of their babies, will be those who require treatment with intravenous antibiotics for at least 36 hours, having been identified as being at risk of having an infection within 12 hours of being born. An infection marker, C-Reactive Protein (CRP) in their blood is measured, and if this remains normal after 18 hours and the baby is suitable for the study, the mother will be given an information leaflet and invitation letter by maternity staff/ ANNPs. Antibiotics will continue to be given to the baby for at least 36- 47 hours until a blood test shows whether they have an infection or not. If they don't have an infection and are healthy, they will be considered for this study.

Both groups of babies are regularly monitored by the staff in the maternity unit to make sure that any problems they have are acted on quickly. Both groups of babies would normally be in hospital for 36- 48 hours for this monitoring.

When the babies in both groups are 48-72 hours old, the ANNPs will ask the mother if she is happy for her baby to have an electrocardiogram (ECG) to look at their heart beat pattern. After consideration time, a consent form is signed, a data collection sheet completed, and the ECG is carried out on the baby. This will happen on the ward so there is minimal disruption to the mother and baby.

The ECG machine used is very accurate so if it shows the heart beat pattern is normal, the parents are told the result and can go home. The ANNPs and Doctors specialising in the care of newborn babies will check the result within 24 hours.

If the ECG machine says the heart beat pattern is not normal, then the baby remains in hospital, whilst the result is checked by the ANNPs and the Doctors specialising in the care of newborn babies, as soon as possible after it is taken. If the heart beat reading is abnormal, the ANNPs and Doctors specialising in the care of newborn babies will talk to the parents about further tests and other monitoring.

If the confirmed ECG result is known before discharge home, the General Practitioner (GP) / Community staff will be told of the study and the result, on the hospital discharge letter the mother takes home for them. If the family have gone home before this happens they will receive a confirmed normal result in the post. The confirmed result will also be added to the electronic hospital records.

In order to give statistically significant results, the study will be carried out over 12 -18 months, and involve 121 babies in each group. After 50 babies have had an ECG, the results will be reviewed to see what results are being seen and to see if the study is following the original plan/ time frame.

A statistician helped to determine how many babies would be needed for the study to show a difference between the two groups. However even if the difference is less than expected, the study may still point to the possibility of an association and provide useful data for future studies.

ELIGIBILITY:
Inclusion Criteria:

* Neonates 37 weeks or more gestation at birth
* Age of parent/ person with parental responsibility being at least 16 years old
* Clinically well parent/ person with parental responsibility
* English Speaking parent/ person with parental responsibility
* Neonate at least 48 hours old

Inclusion criteria for case group participants only:

* Maternal SSRI use at any point in pregnancy

Inclusion criteria for control group participants only:

* Neonate highlighted as at risk of infection and:-

  * antibiotic therapy at less than 12 hours old;
  * CRP x 2 <10mg/l;
  * negative blood culture at 36-47 hours of age (depending on when antibiotic therapy was . commenced)
  * clinically well on examination by ANNP/ Medical team.

Exclusion Criteria:

* Neonates less than 37 weeks gestation at birth
* Age of parent/ person with parental responsibility under 16 years old
* Neonate who is clinically unwell with risk of infection on examination
* Neonate with CRP greater than 10 mg/l
* Neonate with positive blood culture
* Neonate less than 48 hours old
* Maternal cocaine misuse
* Maternal methadone use
* Maternal use of other antidepressants
* Known maternal or fetal structural cardiac abnormality
* Neonate with heart murmur at the time of the planned ECG
* Neonate presenting with congenital abnormality with a high incidence of associated cardiac malformations . . in current pregnancy (e.g., Trisomy 21)

Exclusion criteria for case group participants only:-

* Neonate highlighted as at risk of infection and requiring antibiotic therapy.

Exclusion criteria for control group participants only:-

* Maternal use of SSRIs in pregnancy

Ages: 2 Days to 3 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 88 (Actual)
Dates: Start 2016-02-18 (Actual); Primary Completion 2017-08-18 (Actual); Study Completion 2017-08-18 (Actual)

PRIMARY OUTCOMES:
QT interval on ECG of 48-72 hours old neonates | 48-72 hours old
  The range of QT intervals for this age group of neonates will be ascertained on ECG. Those outside the accepted norm of 2 deviations from the mean (>440msecs) will be highlighted as prolonged.

SECONDARY OUTCOMES:
SSRIs taken antenatally as stated on the data collection sheet. | 48 -72 hours postpartum
  The range of SSRIs taken in pregnancy locally will be extracted from the data collection sheet.
Gestation at which SSRIs were taken as stated on the data collection sheet. | 48 -72 hours postpartum
  The timeline for SSRI use in pregnancy locally will be extracted from the data collection.
Wellbeing as stated in hospital record at 6 months of age if prolonged QT interval on ECG at 48- 72 hours of age. | 6 months old
  Mortality and morbidity assessment by reviewing the electronic patient record at 6 months of age of only those neonates who presented with early prolongation of the QT interval.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Southampton, Southampton, Hampshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
Not personal details but details in questionnaire will be included in articles as a group. Undecided whether it will draw on individual aspects

REFERENCES:
- [Background] Dubnov-Raz G, Juurlink DN, Fogelman R, Merlob P, Ito S, Koren G, Finkelstein Y. Antenatal use of selective serotonin-reuptake inhibitors and QT interval prolongation in newborns. Pediatrics. 2008 Sep;122(3):e710-5. doi: 10.1542/peds.2008-0658. PMID 18762507
- [Background] Lattimore KA, Donn SM, Kaciroti N, Kemper AR, Neal CR Jr, Vazquez DM. Selective serotonin reuptake inhibitor (SSRI) use during pregnancy and effects on the fetus and newborn: a meta-analysis. J Perinatol. 2005 Sep;25(9):595-604. doi: 10.1038/sj.jp.7211352. PMID 16015372
- [Background] Tuccori M, Testi A, Antonioli L, Fornai M, Montagnani S, Ghisu N, Colucci R, Corona T, Blandizzi C, Del Tacca M. Safety concerns associated with the use of serotonin reuptake inhibitors and other serotonergic/noradrenergic antidepressants during pregnancy: a review. Clin Ther. 2009 Jun;31 Pt 1:1426-53. doi: 10.1016/j.clinthera.2009.07.009. PMID 19698902
- [Background] Udechuku A, Nguyen T, Hill R, Szego K. Antidepressants in pregnancy: a systematic review. Aust N Z J Psychiatry. 2010 Nov;44(11):978-96. doi: 10.3109/00048674.2010.507543. PMID 21034181